CLINICAL TRIAL: NCT05896059
Title: A Phase II, Open-Label, Single-Arm, Prospective Clinical Study to Investigate the Efficacy and Safety of Tislelizumab Combined With Anlotinib as Maintenance Therapy Following Tislelizumab and Chemotherapy for Treatment Naïve Extensive Stage Small Cell Lung Cancer
Brief Title: A Study to Investigate the Efficacy and Safety of Tislelizumab Combined With Anlotinib as Maintenance Therapy for ES-SCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Fan Yun, MD, Director of department, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2022]-12-23
Record Dates: First submitted 2023-05-24; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Extensive Stage Small Cell Lung Cancer
MeSH Terms: interventions — tislelizumab; anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab combined with Anlotinib (Experimental)
  Interventions: Drug: Tislelizumab; Drug: Anlotinib

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab，200mg，D1, intravenous，Q3W；
Drug: Anlotinib — Anlotinib，12mg，oral administration，QD.

SUMMARY:
This is an open-label, single-arm, prospective phase 2 study, evaluating the efficacy and safety of tislelizumab combined with Anlotinib as maintenance therapy following tislelizumab and chemotherapy for treatment naïve extensive stage small cell lung cancer.

DETAILED DESCRIPTION:
The study included screening period, treatment period (including induction and maintenance), safety follow-up and survival follow-up periods.

Induction treatment will be administered on a Q3W cycle for 4 cycles. Following induction treatment, patients who have received 4 cycles of tislelizumab and platinum-based chemotherapy and meet the following criteria will enter a maintenance treatment phase with tislelizumab and Anlotinib.

Patients have an ongoing response per RECIST v1.1 criteria of SD or better assessed by the investigator according to RECIST v1.1（Patients will be eligible to enter maintenance phase if chemotherapy interruption due to toxicity, but at least 3 cycles of tislelizumab combined with chemotherapy are completed and assessed as CR, PR or SD according to RECISTv1.1 criteria）.

Excluded patients with central cavitary ES-SCLC, or tumor invading or adjacent to large vessels as shown by imaging, and likely to invade large vessels and cause fatal bleeding assessed by the investigator.

During the maintenance treatment period prophylactic cranial irradiation (PCI) is permitted as per local standard of care.

Treatment may continue until 1) disease progression as assessed by the investigator per RECIST v1.1, 2) loss of clinical benefit as assessed by the investigator, 3) unacceptable toxicity, or 4) withdrawal of informed consent, whichever occurs first, 5) study treatment duration reached 2 years (including induction and maintenance period).

Per investigator's discretion, patients who may continue to benefit from study treatment after progressive disease must meet the following criteria in order to be treated and documented in the study records:

Absence of symptoms and signs indicating clinically significant progression of disease and absence of worsening of laboratory values indicating disease progression.

Stable ECOG performance status ≤ 1 Absence of rapid progression of disease or of progressive tumor at critical anatomical sites (eg,cord compression) that requires urgent alternative medical intervention Investigators must obtain written informed consent for treatment beyond radiologic disease.

Study treatment will be administered for up to 2 years (including induction and mantenance period).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed ES-SCLC, defined by the American Joint Committee on Cancer (AJCC) 8th edition or the Veterans Administration Lung Study Group (VALG) staging system.
2. No prior treatment for ES-SCLC. (Patients who have received prior chemoradiotherapy for limited-stage SCLC must have been treated with curative intent and experienced a treatment-free interval of ≥ 6 months between the completion of chemotherapy, radiotherapy, or chemoradiotherapy and diagnosis of ES-SCLC).
3. ECOG performance status ≤ 1.
4. Life expectancy ≥ 3 months.

   Adequate organ function as indicated by the following laboratory values (obtained ≤ 7 days before first dose):
5. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelets ≥ 100 × 109/L，hemoglobin ≥ 90 g/L.
6. International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 x upper limit of normal (ULN).
7. Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN.
8. Serum total bilirubin ≤ 1.5 x ULN.
9. Aspartate and alanine aminotransferase (AST and ALT) ≤ 2.5 x ULN, or AST and ALT ≤ 5 x ULN for patients with liver metastases.
10. Serum albumin (ALB) ≥ 25g/L.
11. Serum creatinine ≤ 1.5 x ULN or estimated glomerular filtration rate (GFR) ≥ 60 mL/min/1.73 m2 by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.
12. Able to provide written informed consent by the patient or by the patient's legally acceptable representative and can understand and agree to comply with the requirements of the study.
13. 18 to 75 years old on the day of signing the informed consent form (ICF).
14. Fertile patients must be willing to use highly effective contraception during the study period and for 120 days after the last dose of tislelizumab.

Exclusion Criteria:

1. Active leptomeningeal disease or uncontrolled, untreated brain metastasis:

   Patients with a history of treated and, at the time of screening, asymptomatic central nervous system (CNS) metastases are eligible if they meet all the following:
   * only supratentorial metastases allowed.
   * No radiotherapy for the central nervous system within 14 days prior to screening.
   * Untreated and Asymptomatic patients with brain metastasis brain metastases can be included in the study after judgment by the investigators, but regular brain imaging examinations of the disease site are required.
2. Received prior therapies targeting PD-1, PD-L1, CTLA-4 or other immune checkpoints.
3. Received prior anti-VEGF or VEGFR TKI agents including but not limited to Anlotinib.
4. Treatment with any approved systemic anti-cancer therapy or systemic immune-stimulatory agents (including but not limited to interferons, interleukin IL-2, and tumor necrosis factor) within 28 days prior to initiation of study treatment.
5. Clinically uncontrolled pleural effusion, ascites, pericardial effusion that requires treatment and may affect study treatment estimated by investigator.
6. History of allergic reactions to any study drugs or any component of the preparation or any component of the container.
7. Patients with untreated chronic hepatitis B (HBV) or chronic HBV carriers whose HBV DNA ≥ 500 IU/mL (2500 copies/mL), patients with active hepatitis C (HCV).
8. Active autoimmune diseases that require treatment and may affect study treatment estimated by investigator.
9. Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or any other immunosuppressive medication≤ 14 days before first dose of study drugs that may affect study treatment estimated by investigator.
10. Severe chronic or active infections requiring systemic antibacterial, antifungal, or antiviral therapy, within 14 days prior to first dose of study drug(s). Note: antiviral therapy is permitted for patients with viral hepatitis.
11. Prior allogeneic stem cell transplantation or organ transplantation.
12. Any of the following cardiovascular risk criteria:

    1. Cardiac chest pain, defined as moderate pain that limits instrumental activities of daily living, ≤ 28 days before first dose of study drugs.
    2. Symptomatic pulmonary embolism ≤ 28 days before first dose of study drugs.
    3. Any history of acute myocardial infarction ≤ 6 months before first dose of study drugs.
    4. Any history of heart failure meeting New York Heart Association Classification III or IV ≤ 6 months before first dose of study drugs.
    5. Any event of ventricular arrhythmia ≥ Grade 2 in severity ≤ 6 months before first dose of study drugs.
    6. Any history of cerebrovascular accident ≤ 6 months before first dose of study drugs.
    7. QTc interval (corrected by Fridericia's method) > 450 msec (for males)/ > 470 msec (for females).

       Note: If QTc interval is > ULN on initial ECG, a follow up ECG will be performed to exclude result.
    8. Current left ventricular ejection fraction (LVEF) < institutional LLN as assessed by echocardiography (ECHO).
    9. Any episode of syncope or seizure ≤ 28 days before the first dose of study drug(s).
13. Inadequately controlled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg).
14. Bleeding or thrombotic disorders or use of anticoagulants such as warfarin or similar agents requiring therapeutic INR monitoring within 6 months before first dose of study drugs, that may affect study treatment estimated by investigator.
15. Regardless of the severity, patients with any signs or medical history of bleeding; within 4 weeks prior to allocation, patients with any bleeding events ≥ CTCAE level 3, unhealed wounds, ulcers, or fractures.
16. Hemoptysis>50ml/d.
17. Inability to swallow capsules or disease significantly affecting gastrointestinal function, such as malabsorption syndrome, resection of the stomach or small bowel, bariatric surgery procedures, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.
18. History of interstitial lung disease, noninfectious pneumonitis or uncontrolled diseases including pulmonary fibrosis, acute lung diseases, etc, that may affect study treatment estimated by investigator.
19. Significant history or clinical manifestation of any organ systems disorder, as determined by the investigator, that may affect study treatment estimated by investigator.
20. Any major surgical procedure requiring general anesthesia ≤ 28 days before initiation of study treatment.
21. Underlying medical conditions (including laboratory abnormalities) or alcohol or drug abuse or dependence that would be unfavorable for the administration of study drug or affect the explanation of drug toxicity or AEs or result in insufficient or might impair compliance with study conduct.
22. Was administered a live vaccine ≤ 4 weeks before screening.
23. A known history of HIV infection.
24. Any active malignancy ≤ 2 years before first dose of study drugs except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated curatively (e.g., resected basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast).
25. Pregnant or breastfeeding woman.
26. Concurrent participation in another clinical study unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
1-year PFS rate assessed by investigator in maintenance phase-patient analysis set per RECIST v1.1. | Start of maintenance therapy until 1-year follow-up
  PFS is defined as the time from the first dose of study drug(s) in maintenance phase to the first occurrence of disease progression as determined by investigator using RECIST v1.1 or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
PFS | up to 2 year
  PFS assessed by investigators per RECIST v1.1 in maintenance phase-patient analysis set and induction phase-patient analysis set, respectively.
OS | up to 2 year
  OS, defined as the time from first dose of study drug(s) to death from any cause, in maintenance phase-patient analysis set and induction phase-patient analysis set, respectively.
ORR | up to 2 year
  ORR, defined as the proportion of patients with partial response or complete response as determined by the investigators based on RECIST v1.1 in maintenance phase-patient analysis set and induction phase-patient analysis set, respectively.
DCR | up to 2 year
  DCR, defined as the proportion of patients achieving complete response (CR), partial response (PR), or stable disease (SD) as determined by the investigators based on RECIST v1.1 in maintenance phase-patient analysis set and induction phase-patient analysis set, respectively.
DOR | up to 2 year
  DOR is defined as the duration from the date of patients achieve CR or PR to the date of PD or death, which occurs first, for patients with an objective response in maintenance phase-patient analysis set and induction phase-patient analysis set, respectively.
TEAE | up to 2 year
  Incidence and severity of treatment-emergent adverse events (TEAEs) graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0, and relevant physical examinations, electrocardiograms (ECGs), and laboratory assessments as needed. The safety and tolerability will be evaluated in maintenance phase and induction phase population respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided